CLINICAL TRIAL: NCT00045942
Title: An Open-label Phase II (Proof of Concept (POC)) Trial of PKC412 Monotherapy in Participants With Acute Myeloid Leukemia (AML) and Participants With High Risk Myelodysplastic Syndrome (MDS) (CPKC412A2104 Core); An Open-label, Randomized Phase II POC Trial in PKC412 in Participants With AML and Participants With High Risk MDS With Either Wild Type or Mutated FLT3 (CPKC412A2104E1); and An Open-label, Randomized Phase 1/II POC Trial in PKC412 in Participants With AML and Participants With High Risk MDS With Either Wild Type or Mutated FLT3 (CPKC412A2104E2)
Brief Title: PKC412 in Participants With Acute Myeloid Leukemia or With Myelodysplastic Syndrome (CPKC412A2104 Core); and PKC412 in Participants With Acute Myeloid Leukemia or With Myelodysplastic Syndrome With Either Wild Type or Mutated FMS-like Tyrosine Kinase 3 (FLT3) (CPKC412A2104E1 and CPKC412A2104E2)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPKC412A2104; NCT00045578 (obsolete NCT alias); NCT00977782 (obsolete NCT alias)
Record Dates: First submitted 2002-09-16; First posted 2002-09-18 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: AML; MDS; high risk myelodysplastic syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Itraconazole; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- PKC412 (Core) (Experimental): Participants received 75 mg PKC412 three time daily (tid) orally on a continuous basis until disease progression or the occurrence of unacceptable treatment related toxicity.
  Interventions: Drug: PKC412
- FLT3 mutated PKC412 100 mg/day (E1) (Experimental): Participants received 50 mg PKC412 twice daily (bid) orally on a continuous basis until disease progression or the occurrence of unacceptable treatment related toxicity.
  Interventions: Drug: PKC412
- FLT3 mutated PKC412 200 mg/day (E1) (Experimental): Participants received 100 mg PKC412 twice daily (bid) orally on a continuous basis until disease progression or the occurrence of unacceptable treatment related toxicity.
  Interventions: Drug: PKC412
- FLT3 wild type PKC412 100 mg/day (E1) (Experimental): Participants received 50 mg PKC412 twice daily (bid) orally on a continuous basis until disease progression or the occurrence of unacceptable treatment related toxicity.
  Interventions: Drug: PKC412
- FLT3 wild type PKC412 200 mg/day (E1) (Experimental): Participants received 100 mg PKC412 twice daily (bid) orally on a continuous basis until disease progression or the occurrence of unacceptable treatment related toxicity.
  Interventions: Drug: PKC412
- FLT3 mutated PKC412 dose escalation (Experimental): Participants were treated with PKC412 orally starting at a dose of 100 mg bid. A dose increase up to 300 mg bid was allowed. Participants were treated until time of disease progression, doubling of the bone marrow blast percentage from baseline, or the occurrence of unacceptable toxicity.
  Interventions: Drug: PKC412
- FLT3 mutated PKC+Itraconazole (E2) (Experimental): Within a cycle of 28 days, participants received a loading dose of PKC412 100 mg bid on days 1-2, followed by PKC412 50 mg bid for 3 weeks from days 3-21. On day 22, itraconazole 100 mg bid was added to the treatment regimen. The combinations of PKC412 and Itraconazole continued until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Itraconazole; Drug: PKC412
- FLT3 wild type PKC412 dose escalation (E2) (Experimental): Participants were treated with PKC412 orally starting at a dose of 100 mg bid. A dose increase up to 300 mg bid was allowed. Participants were treated until time of disease progression, doubling of the bone marrow blast percentage from baseline, or the occurrence of unacceptable toxicity.
  Interventions: Drug: PKC412
- FLT3 wild type PKC+Itraconazole (E2) (Experimental): Within a cycle of 28 days, participants received a loading dose of PKC412 100 mg bid on days 1-2, followed by PKC412 50 mg bid for 3 weeks from days 3-21. On day 22, itraconazole 100 mg bid was added to the treatment regimen. The combinations of PKC412 and Itraconazole continued until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Itraconazole; Drug: PKC412

INTERVENTIONS:
Drug: Itraconazole — Itraconazole was commercially available.
  Arms: FLT3 mutated PKC+Itraconazole (E2); FLT3 wild type PKC+Itraconazole (E2)
Drug: PKC412 — PKC412 was supplied as soft gelatin capsules containing 25 mg PKC412.
  Other Names: Midostaurin

SUMMARY:
CPKC412A2104 core had a 2 stage design. In stage 1, eight participants were treated. If at least one participant showed a clinical response, four more participants were recruited to stage 2. The trial was to be stopped if no participants showed a response in stage 1. POC was achieved if at least 2 participants out of 12 responded. In PKC412A2104E1, participants with AML or high risk MDS with wild-type or mutant FTL3 who had not previously received a FLT3 inhibitor were randomized to receive continuous twice daily oral doses of either 50 or 100 mg midostaurin in 1 28-day cycle regimen. Participants were to be treated until disease progression or the occurrence of unacceptable treatment-related toxicity. PKC412A2104 E2 contained 2 dosing regimens: 1) intra-participant midostaurin dose escalation and 2) midostaurin with itraconazole in participants with AML and high risk MDS irrespective of FLT3 status. Eligible participants were alternately assigned to the regimens. At the Investigator's discretion, intra-participant dose escalation was allowed for any previously enrolled CPKC412A2104E1 participant receiving midostaurin at the time of the approval of amendment 4. Participants were treated until the time of disease progression.

ELIGIBILITY:
Inclusion criteria:

1. Patients:

   with AML who are not candidates for myelosuppressive chemotherapy or with AML who have relapsed disease or are refractory to standard therapy and not likely to require cytoreductive therapy within one month or with MDS subtypes refractory anemia with excess blasts (RAEB), RAEB in transformation (RAEB-T) or chronic myelomonocytic leukemia (CMML).
2. Patients with a relevant FLT3-ITD mutation or D835Y point mutation
3. Patients at least 18 years or older
4. Patients with WHO performance status of 0 to 2 with a life expectancy of at least 3 months
5. Patients must not be treated within 4 weeks after any prior therapy
6. Written informed consent obtained according to local guidelines

Exclusion criteria:

Patients meeting any of the following criteria during screening will be excluded from entry into the study:

1. Patients who had prior allogeneic, syngeneic, or autologous bone marrow transplant or stem cell transplant less than 2 months previously.
2. Female patients who are pregnant or breast feeding, or adults of childbearing age not employing an effective method of birth control.
3. Concurrent severe and/or uncontrolled medical or psychiatric condition which may interfere with the completion of the study.
4. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PKC412.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2002-01-30 (Actual); Primary Completion 2008-03-27 (Actual); Study Completion 2008-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - UCLA Medical Center, Los Angeles, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - New York Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In PKC412A2104 (Core), FLT3 mutated participants with AML or MDS received open-label PKC412. In PKC412A2104E1, FLT3 mutated participants and FLT3 wild type participants were randomized to receive either PKC412 50 mg bid or PKC412 100 mg bid.
Pre-assignment Details: In PKC412A2104E2, participants were alternately assigned to the regimens, beginning with the first enrolled into the intra-patient dose escalation arm and the next enrolled into the PKC412 + itraconazole arm. Of the 16 participants enrolled in the PKC412 dose escalation arm, 14 were newly enrolled, and 2 were transitioned from PKC412A2104E1.
Groups:
- PKC412 in FLT3 Mutated Participants (Core): Participants received 75 mg PKC412 three time daily (tid) orally on a continuous basis until disease progression or the occurrence of unacceptable treatment related toxicity.
- FLT3 Mutated PKC412 Dose Escalation (E2); FLT3 Wild Type PKC412 Dose Escalation (E2): Participants were treated with PKC412 orally starting at a dose of 100 mg bid. A dose increase up to 300 mg bid was allowed. Participants were treated until time of disease progression, doubling of the bone marrow blast percentage from baseline, or the occurrence of unacceptable toxicity.
Period: PKC412A2104 (Core)
Arm/Group | PKC412 in FLT3 Mutated Participants (Core) | FLT3 Mutated PKC412 100 mg/Day (E1) | FLT3 Mutated PKC412 200 mg/Day (E1) | FLT3 Wild Type PKC412 100 mg/Day (E1) | FLT3 Wild Type PKC412 200 mg/Day (E1) | FLT3 Mutated PKC412 Dose Escalation (E2) | FLT3 Mutated PKC+Itraconazole (E2) | FLT3 Wild Type PKC412 Dose Escalation (E2) | FLT3 Wild Type PKC+Itraconazole (E2)
Started | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Core Primary Efficacy | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: PKC412A2104E1
Arm/Group | PKC412 in FLT3 Mutated Participants (Core) | FLT3 Mutated PKC412 100 mg/Day (E1) | FLT3 Mutated PKC412 200 mg/Day (E1) | FLT3 Wild Type PKC412 100 mg/Day (E1) | FLT3 Wild Type PKC412 200 mg/Day (E1) | FLT3 Mutated PKC412 Dose Escalation (E2) | FLT3 Mutated PKC+Itraconazole (E2) | FLT3 Wild Type PKC412 Dose Escalation (E2) | FLT3 Wild Type PKC+Itraconazole (E2)
Started | 0 | 18 | 17 | 33 | 27 | 0 | 0 | 0 | 0
Primary Efficacy | 0 | 18 | 17 | 32 | 25 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 18 | 17 | 33 | 27 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 5 | 2 | 0 | 0 | 0 | 0
Not completed — Condition no longer requires study drug | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 11 | 11 | 23 | 17 | 0 | 0 | 0 | 0
Not completed — Abnormal laboratory value | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 3 | 6 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 4 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Enrolled into PKC412A2104E2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: PKC412A2104E2
Arm/Group | PKC412 in FLT3 Mutated Participants (Core) | FLT3 Mutated PKC412 100 mg/Day (E1) | FLT3 Mutated PKC412 200 mg/Day (E1) | FLT3 Wild Type PKC412 100 mg/Day (E1) | FLT3 Wild Type PKC412 200 mg/Day (E1) | FLT3 Mutated PKC412 Dose Escalation (E2) | FLT3 Mutated PKC+Itraconazole (E2) | FLT3 Wild Type PKC412 Dose Escalation (E2) | FLT3 Wild Type PKC+Itraconazole (E2)
Started | 0 | 0 | 0 | 0 | 0 | 9 | 7 | 7 | 6
Primary Efficacy | 0 | 0 | 0 | 0 | 0 | 9 | 7 | 7 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 9 | 7 | 7 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline characteristics for PKC412A2104E2 do not include data for the 2 patients who transferred from CPKC412A2104E1 since the data for these 2 patients are included under CPKC412A2104E1.
Groups:
- Total: Total of all reporting groups
Arm/Group | PKC412 in FLT3 Mutated Participants (Core) | FLT3 Mutated PKC412 100 mg/Day (E1) | FLT3 Mutated PKC412 200 mg/Day (E1) | FLT3 Wild Type PKC412 100 mg/Day (E1) | FLT3 Wild Type PKC412 200 mg/Day (E1) | FLT3 Mutated PKC412 Dose Escalation (E2) | FLT3 Mutated PKC+Itraconazole (E2) | FLT3 Wild Type PKC412 Dose Escalation (E2) | FLT3 Wild Type PKC+Itraconazole (E2) | Total
Number analyzed (Participants) | 20 | 18 | 17 | 33 | 27 | 8 | 7 | 6 | 6 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 8 | 7 | 8 | 6 | 5 | 0 | 0 | 56
  >=65 years | 9 | 7 | 9 | 26 | 19 | 2 | 2 | 6 | 6 | 86
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 9 | 17 | 15 | 3 | 3 | 4 | 4 | 66
  Male | 14 | 13 | 8 | 16 | 12 | 5 | 4 | 2 | 2 | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Best Clinical Response (Core)
Description: Best clinical response was defined as complete response (CR) or partial response (PR), according to NCI definitions for AML and the guidelines for defining responses in MDS.
Time Frame: from date of first patient first visit (FPFV), 29-Jan-2002, to date of last participant last visit (LPLV), 04-Sep-2003
Population: Core primary efficacy population: The core primary efficacy population included all participants who were randomized.
Measure: Number; unit: Participants
Arm/Group | PKC412 in FLT3 Mutated Participants (Core)
Number analyzed (Participants) | 20
Participants | 0

2. Primary Outcome: Percent Decrease in Phospho-FLT3 Compared to Baseline (Core)
Time Frame: days 1, 28
Population: This outcome measure was not analyzed. Assessment of FLT3 autophosphorylation in leukemic blasts was not possible at the planned time points because the blast reduction was rapid and occurred during the first week in some participants. Thus, by Day 28, the blast count in some participants were too low for autophosphorylation to be measured.
Arm/Group | PKC412 in FLT3 Mutated Participants (Core)
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants With Overall Clinical Response (E1)
Description: Overall clinical response was defined as CR, PR, minor response (MR) or blast response (BR). CR and PR was defined according to NCI definitions, and MR and BR was defined according to the guidelines for defining hematologic improvement in MDS.
Time Frame: from date of FPFV, 27-Mar-2003, to date of LPLV, 06-Sep-2004
Population: E1 primary efficacy population: all participants who received at least one dose of study medication, completed at least 8 days of therapy within Cycle 1 unless discontinued due to progressive disease and/or death due to any cause, and who were not considered to be associated with a protocol violation that was exclusionary from the population.
Measure: Number; unit: Participants
Arm/Group | FLT3 Mutated PKC412 100 mg/Day (E1) | FLT3 Mutated PKC412 200 mg/Day (E1) | FLT3 Wild Type PKC412 100 mg/Day (E1) | FLT3 Wild Type PKC412 200 mg/Day (E1)
Number analyzed (Participants) | 18 | 17 | 32 | 25
Participants
  Complete response | 0 | 0 | 0 | 0
  Partial response | 0 | 1 | 0 | 0
  Minor response | 1 | 0 | 6 | 3
  Blast response | 11 | 12 | 15 | 8
  Overall response | 12 | 13 | 21 | 11

4. Primary Outcome: Percent Decrease in Phospho-FLT3 Compared to Baseline (E1)
Time Frame: days 1, 28
Population: The analyses for this outcome measure were not performed due to technical challenges in measuring phosphorylated FLT3 in patient blast samples in an ex vivo setting.
Arm/Group | FLT3 Mutated PKC412 100 mg/Day (E1) | FLT3 Mutated PKC412 200 mg/Day (E1) | FLT3 Wild Type PKC412 100 mg/Day (E1) | FLT3 Wild Type PKC412 200 mg/Day (E1)
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Primary Outcome: Percent Decrease in Phospho-FLT3 Compared to Baseline (E2)
Time Frame: Days 1, 28
Population: as for outcome 4
Arm/Group | FLT3 Mutated PKC412 Dose Escalation (E2) | FLT3 Mutated PKC+Itraconazole (E2) | FLT3 Wild Type PKC412 Dose Escalation (E2) | FLT3 Wild Type PKC+Itraconazole (E2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau) for PKC412 Plasma in the PKC + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for pharmacokinetic (PK) analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: The pharmacokinetic (PK) population in the midostaurin + itraconazole FLT3 mutated and FLT3 wild-type combined arms, which consisted of 10 participants, was considered for the analysis. For each time point, participants of the PK analysis set with non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/ml
Groups:
- FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined: Within a cycle of 28 days, participants received a loading dose of PKC412 100 mg bid on days 1-2, followed by PKC412 50 mg bid for 3 weeks from days 3-21. On day 22, itraconazole 100 mg bid was added to the treatment regimen. The combinations of PKC412 and Itraconazole continued until disease progression, unacceptable toxicity, or withdrawal of consent.
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 10
h*ng/ml
  Cycle 1, day 21 (n=9) | 22261.53 (11984.6)
  Cycle 1, day 22 (n=10) | 37578.85 (44330.7)
  Cycle 1, day 28 (n=7) | 35630.45 (23993.2)

7. Primary Outcome: Observed Maximum Plasma Concentration Following Drug Administration at Steady State (Cmax) for PKC412 in the PKC + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for pharmacokinetic (PK) analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 10
ng/ml
  Cycle 1 , day 21 (n=10) | 3945.00 (4440.238)
  Cycle 1, day 22 (n=10) | 3968.70 (4047.498)
  Cycle 1, day 28 (n=8) | 3931.25 (2638.135)

8. Primary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax) for PKC412 in the PKC412 + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for PK analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 10
hour
  Cycle 1, day 21 (n=10) | 1.6 [1.0 to 8.1]
  Cycle 1, day 22 (n=10) | 1.9 [1.2 to 4.7]
  Cycle 1, day 28 (n=8) | 2.2 [0.0 to 3.3]

9. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) for PKC412 in the PKC412 + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for PK analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 10
h*ng/ml
  Cycle 1, day 21 (n=10) | 32120.58 (35792.2)
  Cycle 1, day 22 (n=10) | 34684.6 (37084.9)
  Cycle 1, day 28, (n=8) | 33020.17 (17206.3)

10. Primary Outcome: Terminal Elimination Half-life (T1/2) for PKC412 in the PKC + Itrconazole Combination Arm (E2)
Description: Blood samples were collected for PK analysis.
Time Frame: Cycle 1: days 21 and 22
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 8
hour
  Cycle 1, day 21 (n=6) | 18.13 (13.505)
  Cycle 1, day 22 (n=8) | 13.23 (6.346)

11. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau) for CGP62221 Plasma in the PKC + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for pharmacokinetic (PK) analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 8
h*ng/ml
  Cycle 1, day 21 (n=8) | 30217.82 (16502.90)
  Cycle 1, day 22 (n=7) | 23824.69 (13300.69)
  Cycle 1, day 28 (n=7) | 31545.54 (12453.16)

12. Primary Outcome: Observed Maximum Plasma Concentration Following Drug Administration at Steady State (Cmax) for CGP62221 in the PKC + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for pharmacokinetic (PK) analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 10
ng/ml
  Cycle 1, day 21 (n=10) | 3259.30 (1747.923)
  Cycle 1, day 22 (n=10) | 3221.40 (1980.217)
  Cycle 1, day 28 (n=8) | 3032.25 (1975.371)

13. Primary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax) for CGP62221 in the PKC412 + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for PK analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 10
hour
  Cycle 1, day 21 (n=10) | 3.7 [0.0 to 10.3]
  Cycle 1, day 22 (n=10) | 2.3 [0.0 to 6.1]
  Cycle 1, day 28 (n=8) | 3.3 [0.0 to 8.5]

14. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) for CGP622221 in the PKC412 + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for PK analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 10
h*ng/ml
  Cycle 1, day 21 (n=10) | 31699.93 (15573.87)
  Cycle 1, day 22 (n=10) | 31182.90 (17380.39)
  Cycle 1, day 28 (n=8) | 26688.60 (10901.40)

15. Primary Outcome: Terminal Elimination Half-life (T1/2) for CGP62221 in the PKC + Itrconazole Combination Arm (E2)
Description: Blood samples were collected for PK analysis.
Time Frame: Cycle 1: day 22,
Population: The pharmacokinetic (PK) population in the midostaurin + itraconazole FLT3 mutated and FLT3 wild-type combined arms, which consisted of 10 participants, was considered for the analysis. For this end point, 4 participants with non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 4
hour | 14.37 (6.743)

16. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau) for CGP52421 Plasma in the PKC + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for pharmacokinetic (PK) analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 9
h*ng/ml
  Cycle 1, day 21 (n=9) | 40258.65 (9747.374)
  Cycle 1, day 22 (n=7) | 42950.76 (8604.972)
  Cycle 1, day 28 (n=7) | 49758.77 (7733.621)

17. Primary Outcome: Observed Maximum Plasma Concentration Following Drug Administration at Steady State (Cmax) for CGP52421 in the PKC + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for pharmacokinetic (PK) analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 10
ng/ml
  Cycle 1, day 21 (n=10) | 4173.00 (985.473)
  Cycle 1, day 22 (n=10) | 4293.00 (1292.380)
  Cycle 1, day 28 (n=8) | 4875.00 (1376.382)

18. Primary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax) for CGP52421 in the PKC412 + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for PK analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 10
hour
  Cycle 1, day 21 (n=10) | 3.5 [0.0 to 6.5]
  Cycle 1, day 22 (n=10) | 2.1 [0.0 to 10.7]
  Cycle 1, day 28 (n=8) | 2.2 [0.0 to 8.3]

19. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) for CGP52421 in the PKC412 + Itraconazole Combination Arm (E2)
Description: Blood samples were collected for PK analysis.
Time Frame: Cycle 1: days 21, 22, 28
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | FLT3 Mutated and FLT3 Wild Type PKC + Itraconazole Combined
Number analyzed (Participants) | 10
h*ng/ml
  Cycle 1, day 21 (n=10) | 38899.84 (7616.481)
  Cycle 1, day 22 (n=10) | 41035.50 (10807.22)
  Cycle 1, day 28 (n=8) | 44447.05 (8906.006)

20. Primary Outcome: Summary of Midostaurin Concentration in the PKC412 Dose Escalation Arms(E2)
Description: Blood samples were collected for analysis.
Time Frame: Cycle 1: days 1, 2 (24 hr post day 1), 3, 8, 15, 16 (24 hr post day 15), 17, 22; Cycle 2: days 1, 2 (24 hr post day 1), 3, 8, 15
Population: The PK analysis set of the FLT3 mutated PKC412 dose escalation and FLT3 wild type PKC412 dose escalation combined arms, which consisted of the 14 newly enrolled participants, was considered for the analysis. For each time point, participants of the PK analysis set with non-missing values were analyzed.
Measure: Median (Full Range); unit: ng/ml
Groups:
- FLT3 Mutated and Wild Type PKC412 Dose Escalation Combined: Participants were treated with PKC412 orally starting at a dose of 100 mg bid. A dose increase up to 300 mg bid was allowed. Participants were treated until time of disease progression, doubling of the bone marrow blast percentage from baseline, or the occurrence of unacceptable toxicity.
Arm/Group | FLT3 Mutated and Wild Type PKC412 Dose Escalation Combined
Number analyzed (Participants) | 12
ng/ml
  Cycle 1, day 1 (=7) | 0 [0 to 0]
  Cycle 1, day 2 (24 hours post day 1) (n=12) | 2565.0 [1170.0 to 7250.0]
  Cycle 1, day 3 (n=12) | 3100.0 [1340.0 to 9080.0]
  Cycle 1, day 8 (n=8) | 1640.0 [1030.0 to 4340.0]
  Cycle 1, day 15 (n=6) | 744.5 [549.0 to 7080.0]
  Cycle 1, day 16 (24 hr post day 15) (n=6) | 836.0 [669.0 to 9120.0]
  Cycle 1, day 17 (n=5) | 800.0 [710.0 to 982.0]
  Cycle 1, day 22 (n=5) | 1410.0 [595.0 to 6270.0]
  Cycle 2, day 1 (n=4) | 772.0 [667.0 to 2670.0]
  Cycle 2, day 2 (24 hr post day 1) (n=4) | 1141.0 [516.0 to 6410.0]
  Cycle 2, day3 (n=4) | 1295.0 [610.0 to 7450.0]
  Cycle 2, day 8 (n=4) | 1210.0 [727.0 to 1420.0]
  Cycle 2, day 15 (n=3) | 834.0 [515.0 to 1000.0]

21. Primary Outcome: Summary of CGP62221 Concentration (E2)
Description: Blood samples were collected for analysis.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Median (Full Range); unit: ng/ml
Arm/Group | FLT3 Mutated and Wild Type PKC412 Dose Escalation Combined
Number analyzed (Participants) | 12
ng/ml
  Cycle 1, day 1 (n=7) | 0 [0 to 0]
  Cycle 1, day 2 (24 hr post day 1) (n=12) | 1320.0 [570.0 to 2720.0]
  Cycle 1, day 3 (n=12) | 2750.0 [1800.0 to 4340.0]
  Cycle 1, day 8 (n=8) | 2380.0 [2000.0 to 7380.0]
  Cycle 1, day 15 (n=6) | 1505.0 [1110.0 to 4630.0]
  Cycle 1, day 16 (24 hr post day 15) (n=6) | 1425.0 [1190.0 to 5390.0]
  Cycle 1, day 17 (n=5) | 1480.0 [1200.0 to 1710.0]
  Cycle 1, day 22 (n=5) | 1520.0 [1410.0 to 3330.0]
  Cycle 2, day 1 (n=4) | 1545.0 [1350.0 to 3210.0]
  Cycle 2, day 2 (24 hr post day 1) (n=4) | 1945.0 [880.0 to 3430.0]
  Cycle 2, day 3 (n=4) | 2070.0 [1260.0 to 3430.0]
  Cycle 2, day 8 (n=4) | 2030.0 [1620.0 to 2360.0]
  Cycle 2, day 15 (n=3) | 1740.0 [1360.0 to 1790.0]

22. Primary Outcome: Summary of CGP52421 Concentration (E2)
Description: Blood samples were collected for analysis.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Median (Full Range); unit: ng/ml
Arm/Group | FLT3 Mutated and Wild Type PKC412 Dose Escalation Combined
Number analyzed (Participants) | 12
ng/ml
  Cycle 1, day 1 (n=7) | 0 [0 to 0]
  Cycle 1, day 2 (24 hr post day 1) (n=12) | 684.0 [0.0 to 1100.0]
  Cycle 1, day 3 (n=12) | 1185.0 [1020.0 to 1860.0]
  Cycle 1, day 8 (n=8) | 2835.0 [2230.0 to 3950.0]
  Cycle 1, day 15 (n=6) | 3845.0 [1810.0 to 6110.0]
  Cycle 1, day 16 (24 hr post day 15) (n=6) | 3830.0 [1830.0 to 6070.0]
  Cycle 1, day 17 (n=5) | 3620.0 [2120.0 to 4560.0]
  Cycle 1, day 22 (n=5) | 4470.0 [1860.0 to 8500.0]
  Cycle 2, day 1 (n=4) | 4915.0 [379.0 to 6590.0]
  Cycle 2, day 2 (24 hr post day 1) (n=4) | 4455.0 [185.0 to 9610.0]
  Cycle 2, day 3 (n=4) | 4470.0 [3150.0 to 5210.0]
  Cycle 2, day 8 (n=4) | 4860.0 [3500.0 to 5570.0]
  Cycle 2, day 15 (n=3) | 4030.0 [3370.0 to 5780.0]

23. Secondary Outcome: Time to Disease Progression (TTP) (Core)
Description: TTP was defined as the time from first dose date to date of disease progression which is identified as study completion date for unsatisfactory treatment effect or date of death from any cause within the 28 day cutoff post treatment.
Time Frame: from date of FPFV, 29-Jan-2002, to date of LPLV, 04-Sep-2003
Population: Core primary efficacy population: The core primary efficacy population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PKC412 in FLT3 Mutated Participants (Core)
Number analyzed (Participants) | 20
days | 63.0 [26.0 to 92.0]

24. Secondary Outcome: Summary of Midostaurin Plasma Concentration (Core)
Description: Blood samples were collected for analysis.
Time Frame: Cycle 1: days 1 (24 hour), 3, 8; Cycle 2: day 1,
Population: The Core PK analysis set, which consisted of 15 participants, was considered for the analysis. For each time point, only participants of the PK set who had non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PKC412 in FLT3 Mutated Participants (Core)
Number analyzed (Participants) | 10
ng/ml
  Cycle 1, day 1(24 hour) (n=10) | 3801.0 (2529.069)
  Cycle 1, day 3 (n=7) | 7152.86 (4254.173)
  Cycle 1, day 8 (n=9) | 5154.44 (5004.511)
  Cycle 2, day 1 (n=6) | 1873.17 (1521.685)

25. Secondary Outcome: Summary of CGP62221 Plasma Concentration (Core)
Description: Blood samples were collected for analysis.
Time Frame: Cycle 1: days 1 (24 hour), 3, 8; Cycle 2: day 1,
Population: The Core PK analysis set, which consisted of 15 participants, were considered for the analysis. For each time point, only participants of the PK set who had non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PKC412 in FLT3 Mutated Participants (Core)
Number analyzed (Participants) | 10
ng/ml
  Cycle 1, day 1 (24 hour) (n=10) | 1636.00 (612.938)
  Cycle 1, day 3 (n=7) | 3143.71 (1147.407)
  Cycle 1, day 8 (n=9) | 4873.33 (3421.593)
  Cycle 2, day 1 (n=6) | 2816.67 (2095.850)

26. Secondary Outcome: Summary of CGP52421 Plasma Concentration (Core)
Description: Blood samples were collected for analysis.
Time Frame: Cycle 1: days 1 (24 hour), 3, 8; Cycle 2: day 1,
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PKC412 in FLT3 Mutated Participants (Core)
Number analyzed (Participants) | 10
ng/ml
  Cycle 1, day 1 (24 hour) (n=10) | 951.70 (297.866)
  Cycle 1, day 3 (n=7) | 1846.57 (657.472)
  Cycle 1, day 8 (n=9) | 6342.22 (2586.440)
  Cycle 2, day 1 (n=6) | 12978.33 (4036.436)

27. Secondary Outcome: Time to Disease Progression (E1)
Description: TTP was defined as the time from the first dose date to the date of disease progression (defined as the study completion date for unsatisfactory treatment effect, date of response assessment of progressive disease, or date of death from any cause). One participant from the wild type 200 mg group did not have any assessment on treatment and therefore was not taken into account for TTP.
Time Frame: from date of FPFV, 27-Mar-2003, to date of LPLV, 06-Sep-2004
Population: Primary efficacy population: defined as all patients who received at least 1 dose of study medication, completed at least eight days of therapy within Cycle 1 unless discontinued due to progressive disease and/or death due to any cause, and who were not considered to be associated with a protocol violation that was exclusionary from the population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FLT3 Mutated PKC412 100 mg/Day (E1) | FLT3 Mutated PKC412 200 mg/Day (E1) | FLT3 Wild Type PKC412 100 mg/Day (E1) | FLT3 Wild Type PKC412 200 mg/Day (E1)
Number analyzed (Participants) | 18 | 17 | 32 | 25
days | 77.0 [36.0 to 109.0] | 50.0 [24.0 to 63.0] | 62.0 [30.0 to 82.0] | 54.0 [29.0 to 84.0]

28. Secondary Outcome: Overall Survival (OS) (E1)
Description: OS was measured from the date of the first dose of treatment to the date of death from any cause or to the last date that the patient was known to be alive (a censored observation).
Time Frame: from date of FPFV, 27-Mar-2003, to date of LPLV, 06-Sep-2004
Population: as for outcome 27
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FLT3 Mutated PKC412 100 mg/Day (E1) | FLT3 Mutated PKC412 200 mg/Day (E1) | FLT3 Wild Type PKC412 100 mg/Day (E1) | FLT3 Wild Type PKC412 200 mg/Day (E1)
Number analyzed (Participants) | 18 | 17 | 32 | 25
days | 99.0 [61.0 to 120.0] | 93.0 [52.0 to 139.0] | 145.0 [75.0 to 257.0] | 159.0 [98.0 to 313.0]

29. Secondary Outcome: Duration of Best Clinical Response (E1)
Description: Duration of best clinical response was measured from the time that the measurement criteria were met for CR, PR, MR (with or without blast reduction) or BR until the first date that recurrent disease was documented (event) or until the date of last follow up.
Time Frame: from date of FPFV, 27-Mar-2003, to date of LPLV, 06-Sep-2004
Population: Responders from the PEP; PEP defined as all patients who received at least 1 dose of study medication, completed at least 8 days of therapy within Cycle 1 unless discontinued due to progressive disease and/or death due to any cause, and who were not considered to be associated with a protocol violation that was exclusionary from the population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FLT3 Mutated PKC412 100 mg/Day (E1) | FLT3 Mutated PKC412 200 mg/Day (E1) | FLT3 Wild Type PKC412 100 mg/Day (E1) | FLT3 Wild Type PKC412 200 mg/Day (E1)
Number analyzed (Participants) | 12 | 13 | 21 | 11
days | 57.0 [8.0 to 86.0] | 29.0 [4.0 to 35.0] | 56.0 [29.0 to 78.0] | 58.0 [9.0 to 192.0]

30. Secondary Outcome: Event-free Survival (E1)
Description: Event-free survival was defined as the time from date of start of treatment to the date of death from any cause, treatment failure or relapse
Time Frame: from date of FPFV, 27-Mar-2003, to date of LPLV, 06-Sep-2004
Population: as for outcome 27
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FLT3 Mutated PKC412 100 mg/Day (E1) | FLT3 Mutated PKC412 200 mg/Day (E1) | FLT3 Wild Type PKC412 100 mg/Day (E1) | FLT3 Wild Type PKC412 200 mg/Day (E1)
Number analyzed (Participants) | 18 | 17 | 32 | 25
days | 60.0 [1.0 to 109.0] | 50.0 [1.0 to 63.0] | 58.0 [1.0 to 82.0] | 1.0 [1.0 to 42.0]

31. Secondary Outcome: Summary of PKC412 Plasma Concentration for 50 mg Twice Daily (Bid) Arm (E1)
Description: Blood samples were collected for analysis.
Time Frame: Cycle 1: days 1 (0h, 4h, 24 h), 3 (0h), 8 (0h); cycle 2: days 1 (0h); cycle 3: day 1 (0h); cycle 4: day 1 (0h)
Population: The PK population of the mutated PKC412 100 mg/day and wild type PKC412 100 mg/day arms combined, which consisted of all participants who provided at least one evaluable PK sample and received at least one dose of study treatment, was considered for the analysis. For each time point, only participants with non-missing values were analyzed..
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- FLT3 Mutated and Wild Type PKC412 100 mg/Day Arms Combined: Participants received 50 mg PKC412 twice daily (bid) orally on a continuous basis until disease progression or the occurrence of unacceptable treatment related toxicity.
Arm/Group | FLT3 Mutated and Wild Type PKC412 100 mg/Day Arms Combined
Number analyzed (Participants) | 43
ng/ml
  Cycle 1, day 1 (0h) (n=43) | 0.000 (0.0000)
  Cycle 1, day 1 (4h) (n=38) | 1198.000 (522.4766)
  Cycle 1, day 1 (24h) (n=39) | 1735.974 (1161.933)
  Cycle 1, day 3 (0h) (n=34) | 2585.471 (1843.852)
  Cycle 1, day 8 (0h) (n=30) | 3576.467 (3263.112)
  Cycle 2, day 1 (0h) (n=22) | 1756.500 (1695.327)
  Cycle 3, day 1 (0h) (n=12) | 2038.417 (2079.252)
  Cycle 4, day 1 (0h) (n=4) | 820.750 (565.0247)

32. Secondary Outcome: Summary of CGP62221 Plasma Concentration for 50 mg Bid Arm (E1)
Description: Blood samples were collected for analysis.
Time Frame: Cycle 1: days 1 (0h, 4h, 24 h), 3 (0h), 8 (0h); cycle 2: days 1 (0h); cycle 3: day 1 (0h); cycle 4: day 1 (0h)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | FLT3 Mutated and Wild Type PKC412 100 mg/Day Arms Combined
Number analyzed (Participants) | 44
ng/ml
  Cycle 1, day 1 (0h) (n=44) | 0.000 (0.0000)
  Cycle 1, day 1 (4h) (n=38) | 367.079 (220.2728)
  Cycle 1, day 1 (24h) (n=39) | 808.182 (375.4818)
  Cycle 1, day 3 (0h) (n=34) | 1400.476 (681.9106)
  Cycle 1, day 8 (0h) (n=30) | 2868.933 (1723.985)
  Cycle 2, day 1 (0h) (n=22) | 1930.000 (1241.980)
  Cycle 3, day 1 (0h) (n=12) | 1971.500 (1519.628)
  Cycle 4, day 1 (0h) (n=4) | 1207.500 (310.5238)

33. Secondary Outcome: Summary of CGP52421 Plasma Concentration for 50 mg Bid Arm (E1)
Description: Blood samples were collected for analysis.
Time Frame: Cycle 1: days 1 (0h, 4h, 24 h), 3 (0h), 8 (0h); cycle 2: days 1 (0h); cycle 3: day 1 (0h); cycle 4: day 1 (0h)
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | FLT3 Mutated and Wild Type PKC412 100 mg/Day Arms Combined
Number analyzed (Participants) | 41
ng/ml
  Cycle 1, day 1 (0h) (n=41) | 0.000 (0.0000)
  Cycle 1, day 1 (4h) (n=38) | 203.013 (121.3817)
  Cycle 1, day 1 (24h) (n=39) | 436.282 (210.1306)
  Day 1, day 3 (0h) (n=34) | 1188.359 (1833.644)
  Cycle 1, day 8 (0h) (n=30) | 2840.833 (1158.132)
  Cycle 2, day 1 (0h) (n=22) | 6467.591 (3434.776)
  Cycle 3, day 1 (0h) (n=12) | 8175.000 (4851.968)
  Cycle 4, day 1 (0h) (n=4) | 6205.000 (1619.084)

34. Secondary Outcome: Summary of PKC412 Plasma Concentration for 100 mg Bid Arm (E1)
Description: Blood samples were collected for analysis.
Time Frame: Cycle 1: days 1 (0h, 4h, 24 h), 3 (0h), 8 (0h); cycle 2: days 1 (0h); cycle 3: day 1 (0h); cycle 4: day 1 (0h); cycle 5: day 1 (0h) and cycle 6: day 1 (0h)
Population: The PK population of the mutated PKC412 200 mg/day and wild type PKC412 200 mg/day arms combined, which consisted of all participants who provided at least one evaluable PK sample and received at least one dose of study treatment, was considered for the analysis. For each time point, only participants with non-missing values were analyzed..
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- FLT3 Mutated and Wild Type PKC412 200 mg/Day: Participants received 100 mg PKC412 twice daily (bid) orally on a continuous basis until disease progression or the occurrence of unacceptable treatment related toxicity.
Arm/Group | FLT3 Mutated and Wild Type PKC412 200 mg/Day
Number analyzed (Participants) | 38
ng/ml
  Cycle 1, day 1 (0h) (n=38) | 0.000 (0.0000)
  Cycle 1, day 1 (4h) (n=34) | 2087.088 (1087.277)
  Cycle 1, day 1 (24h) (n=36) | 2849.731 (2150.176)
  Cycle 1, day 3 (0h) (n=29) | 3756.483 (2549.759)
  Cycle 1, day 8 (0h) (n=24) | 4447.583 (4233.285)
  Cycle 2, day 1 (0h) (n=15) | 1226.333 (894.1562)
  Cycle 3, day 2 (0h) (n=6) | 754.500 (264.6860)
  Cycle 4, day 1 (0h) (n=6) | 1187.167 (1026.004)
  Cycle 5, day 1 (0h) (n=4) | 572.250 (314.7405)
  Cycle 6, day 1 (0h) (n=4) | 1433.250 (1670.029)

35. Secondary Outcome: Summary of CGP62221 Plasma Concentration for 100 mg Bid Arm (E1)
Description: Blood samples were collected for analysis.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | FLT3 Mutated and Wild Type PKC412 200 mg/Day
Number analyzed (Participants) | 39
ng/ml
  Cycle 1, day 1 (0h) (n=39) | 0.000 (0.0000)
  Cycle 1, day 1 (4h) (n=34) | 471.635 (342.7850)
  Cycle 1, day 1 (24h) (n=36) | 1134.764 (655.1779)
  Cycle 1, day 3 (0h) (n=29) | 1944.069 (1049.770)
  Cycle 1, day 8 (0h) (n=24) | 2898.708 (1876.446)
  Cycle 2, day 1 (0h) (n=15) | 1828.667 (650.1524)
  Cycle 3, day 2 (0h) (n=6) | 1258.333 (289.0271)
  Cycle 4, day 1 (0h) (n=6) | 1602.950 (1071.167)
  Cycle 5, day 1 (0h) (n4) | 1111.250 (357.8728)
  Cycle 6, day 1 (0h) (n=4) | 1662.500 (864.4603)

36. Secondary Outcome: Summary of CGP52421 Plasma Concentration for 100 mg Bid Arm (E1)
Description: Blood samples were collected for analysis.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | FLT3 Mutated and Wild Type PKC412 200 mg/Day
Number analyzed (Participants) | 38
ng/ml
  Cycle 1, day 1 (0h) (n=38) | 0.000 (0.0000)
  Cycle 1, day 1 (4h) (n=34) | 257.391 (148.6420)
  Cycle 1, day 1 (24h) (n=36) | 666.194 (313.5770)
  Cycle 1, day 3 (0h) (n=29) | 1394.062 (653.2943)
  Cycle 1, day 8 (0h) (n=24) | 4447.500 (1359.192)
  Cycle 2, day 1 (0h) (n=15) | 9196.667 (3248.590)
  Cycle 3, day 2 (0h) (n=6) | 8811.667 (3376.172)
  Cycle 4, day 1 (0h) (n=6) | 6266.667 (3895.452)
  Cycle 5, day 1 (0h) (n4) | 7845.000 (4078.313)
  Cycle 6, day 1 (0h) (n=4) | 8710.000 (4890.774)

37. Secondary Outcome: Best Clinical Response (E2)
Description: Best clinical response was defined as CR, PR, MR, MR+BR, or BR . CR and PR was defined according to NCI definitions, and MR and BR was defined according to the guidelines for defining hematologic improvement in MDS.
Time Frame: date of FPFV, 21-Aug-2003, to date of LPLV, 27-Mar-2008
Population: The primary efficacy population, which included all participants, who received at least one dose of study drug and who completed at least 8 days of treatment in Cycle 1, unless they discontinued due to progressive disease and/or death due to any cause, and who did not experience any protocol violations, was analyzed..
Measure: Number; unit: Participants
Arm/Group | FLT3 Mutated PKC412 Dose Escalation (E2) | FLT3 Mutated PKC+Itraconazole (E2) | FLT3 Wild Type PKC412 Dose Escalation (E2) | FLT3 Wild Type PKC+Itraconazole (E2)
Number analyzed (Participants) | 9 | 7 | 7 | 6
Participants
  Complete response | 0 | 0 | 0 | 1
  Partial response | 0 | 0 | 0 | 0
  Minor response | 0 | 0 | 0 | 1
  Minor response and blast response | 1 | 0 | 2 | 1
  Blast response | 4 | 0 | 0 | 1
  Best clinical response | 5 | 0 | 2 | 4

38. Secondary Outcome: Time to Disease Progression (E2)
Description: TTP was defined as the time from the first dose date to the date of disease progression, which was defined as the study completion date for unsatisfactory treatment effect, the date of response assessment of progressive disease, or the date of death from any cause
Time Frame: date of FPFV, 21-Aug-2003, to date of LPLV, 27-Mar-2008
Population: as for outcome 37
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FLT3 Mutated PKC412 Dose Escalation (E2) | FLT3 Mutated PKC+Itraconazole (E2) | FLT3 Wild Type PKC412 Dose Escalation (E2) | FLT3 Wild Type PKC+Itraconazole (E2)
Number analyzed (Participants) | 9 | 7 | 7 | 6
days | 49.0 [11.0 to 222.0] | 26.0 [12.0 to 50.0] | 169.0 [113.0 to 370.0] | 78.0 [29.0 to 1348.0]

39. Secondary Outcome: Overall Survival (E2)
Description: OS was measured from the date of the first dose of treatment to the date of death from any cause or the last date the patient was known to be alive (censored observation)
Time Frame: date of FPFV, 21-Aug-2003, to date of LPLV, 27-Mar-2008
Population: as for outcome 37
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | FLT3 Mutated PKC412 Dose Escalation (E2) | FLT3 Mutated PKC+Itraconazole (E2) | FLT3 Wild Type PKC412 Dose Escalation (E2) | FLT3 Wild Type PKC+Itraconazole (E2)
Number analyzed (Participants) | 9 | 7 | 7 | 6
days | 116.0 [11.0 to 222.0] | 75.0 [26.0 to 194.0] | 372.0 [276.0 to NA] — The upper 95% confidence interval could not be calculated. | 220.0 [64.0 to NA] — The upper 95% confidence interval could not be calculated.

ADVERSE EVENTS:
Groups:
- PKC412 Core: Participants received 75 mg PKC412 three time daily (tid) orally on a continuous basis until disease progression or the occurrence of unacceptable treatment related toxicity.
Arm/Group | PKC412 Core | FLT3 Mutated PKC412 100 mg/Day (E1) | FLT3 Mutated PKC412 200 mg/Day (E1) | FLT3 Wild Type PKC412 100 mg/Day (E1) | FLT3 Wild Type PKC412 200 mg/Day (E1) | FLT3 Mutated PKC412 Dose Escalation (E2) | FLT3 Mutated PKC+Itraconazole (E2) | FLT3 Wild Type PKC412 Dose Escalation (E2) | FLT3 Wild Type PKC+Itraconazole (E2)
Serious Adverse Events (participants affected / at risk) | 12/20 | 16/18 | 14/17 | 22/33 | 19/27 | 7/9 | 6/7 | 5/7 | 3/6
Other Adverse Events (participants affected / at risk) | 20/20 | 17/18 | 16/17 | 32/33 | 27/27 | 9/9 | 6/7 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PKC412 Core (N=20) | FLT3 Mutated PKC412 100 mg/Day (E1) (N=18) | FLT3 Mutated PKC412 200 mg/Day (E1) (N=17) | FLT3 Wild Type PKC412 100 mg/Day (E1) (N=33) | FLT3 Wild Type PKC412 200 mg/Day (E1) (N=27) | FLT3 Mutated PKC412 Dose Escalation (E2) (N=9) | FLT3 Mutated PKC+Itraconazole (E2) (N=7) | FLT3 Wild Type PKC412 Dose Escalation (E2) (N=7) | FLT3 Wild Type PKC+Itraconazole (E2) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 1 | 0
Anaemia NOS (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 3 | 9 | 5 | 1 | 0 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 3 | 3 | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Aplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Intestinal prolapse (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Polyp colorectal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Drug interaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Injection site cellulitis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Performance status decreased (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 1 | 5 | 6 | 4 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular damage (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchopneumonia NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candida sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Catheter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Central line infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Perianal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 5 | 1 | 9 | 3 | 1 | 0 | 1 | 0
Pneumonia NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 4 | 1 | 1 | 0 | 0
Sepsis NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue infection NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Thrombophlebitis septic (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Bacteria stool identified (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blast cell count increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 0
Blood amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Culture urine positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibrinolysis increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gram stain positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Troponin NOS (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone infarction (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukaemic infiltration pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukostasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asterixis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolic encephalopathy NOS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tonic clonic movements (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 2 | 2 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Maxillary sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septal panniculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria NOS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Hypotension NOS (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Venous stasis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PKC412 Core (N=20) | FLT3 Mutated PKC412 100 mg/Day (E1) (N=18) | FLT3 Mutated PKC412 200 mg/Day (E1) (N=17) | FLT3 Wild Type PKC412 100 mg/Day (E1) (N=33) | FLT3 Wild Type PKC412 200 mg/Day (E1) (N=27) | FLT3 Mutated PKC412 Dose Escalation (E2) (N=9) | FLT3 Mutated PKC+Itraconazole (E2) (N=7) | FLT3 Wild Type PKC412 Dose Escalation (E2) (N=7) | FLT3 Wild Type PKC+Itraconazole (E2) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 7 | 3 | 3 | 0 | 4 | 4
Anaemia NOS (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 3 | 0 | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 2
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 5 | 0 | 4 | 1 | 2 | 0 | 2 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 5 | 1 | 4 | 4 | 0 | 1 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia NOS (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 2 | 0 | 1 | 3 | 0 | 0 | 0
Tachycardia NOS (Cardiac disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Mastoid disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hyperaldosteronism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 2 | 0 | 6 | 3 | 0 | 3 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 5 | 3 | 8 | 1 | 2 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 8 | 12 | 15 | 5 | 3 | 4 | 3
Diarrhoea NOS (Gastrointestinal disorders) | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0
Gastric dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 5 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Loose stools (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 14 | 11 | 9 | 19 | 16 | 3 | 3 | 5 | 6
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal petechiae (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Perianal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Saliva altered (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Tongue blistering (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 12 | 9 | 13 | 12 | 4 | 2 | 3 | 4
Vomiting NOS (Gastrointestinal disorders) | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 5 | 3 | 6 | 4 | 0 | 0 | 2 | 2
Catheter site erythema (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 2 | 3 | 2 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 2 | 1 | 1 | 2 | 2 | 1 | 1 | 1
Fatigue (General disorders) | 8 | 7 | 6 | 12 | 8 | 3 | 1 | 4 | 2
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 3 | 1 | 2 | 1 | 1 | 0 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 2 | 3 | 1 | 0 | 1 | 0
Oedema NOS (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 8 | 3 | 4 | 8 | 6 | 1 | 1 | 1 | 1
Pain (General disorders) | 0 | 2 | 1 | 5 | 2 | 2 | 0 | 0 | 1
Pain NOS (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 7 | 7 | 5 | 7 | 5 | 4 | 1 | 1 | 2
Rigors (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Submandibular mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal NOS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ano-rectal infection bacterial NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Candidal infection NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Carbuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes viral infection NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 3 | 2 | 1 | 1 | 0 | 0 | 1
Puncture site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1
Upper respiratory tract infection NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 3 | 4 | 1 | 0 | 0 | 1
Vaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood blister (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 4 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury NOS (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 4 | 0 | 3 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 4 | 0 | 3 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 2 | 0 | 3 | 0 | 0 | 1 | 0
Blood amylase increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 3 | 3 | 1 | 1 | 1 | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood in stool (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur NOS (Investigations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spleen palpable (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 3 | 2 | 5 | 4 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 2 | 4 | 0 | 1 | 3 | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1 | 2 | 0 | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 7 | 6 | 8 | 3 | 3 | 1 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 4 | 4 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4 | 3 | 3 | 1 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 3 | 2 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 3 | 3 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 3 | 0 | 1 | 2 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brain mass (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 2 | 7 | 0 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 7 | 5 | 2 | 4 | 5 | 3 | 3 | 3 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Postictal state (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 2 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 3 | 1 | 3 | 3 | 1 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 0 | 2 | 3 | 0 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Hallucination NOS (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 2 | 3 | 4 | 2 | 2 | 0 | 3
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breath sounds decreased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 4 | 6 | 3 | 2 | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 2 | 8 | 8 | 2 | 3 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 4 | 1 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1 | 4 | 1 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lung infiltration NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 4 | 2 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary oedema NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillar ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 1 | 2 | 0 | 2 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 3 | 2 | 1 | 0 | 3 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 2 | 2 | 1 | 0 | 1 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura NOS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 5 | 2 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion NOS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria NOS (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 1
Haematoma NOS (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 2 | 3 | 2 | 1 | 1 | 2 | 0 | 0
Hypotension NOS (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Petechiae (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.